CLINICAL TRIAL: NCT03118921
Title: Body Image Disorder in Anorexia Nervosa and Virtual Reality
Acronym: REVAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: suggestion of an accentuation of the bias of overestimating the silhouette in one of the avatar exposure modalities in virtual reality
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: REVAM
Record Dates: First submitted 2017-04-03; First posted 2017-04-18 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Anorexia
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental): The first session aims to present the virtual reality material that will be used. The second session will take place 2 weeks after the first session and will consist of the use of the immersion software
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — The first session aims to present the virtual reality material that will be used. The second session will take place 2 weeks after the first session and will consist of the use of the immersion software.

SUMMARY:
Evaluation of the tolerance and acceptability of the virtual representation of its body image.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged between 16 and 40
* Post-puberty
* Pure restrictive anorexia nervosa, diagnosis by the DSM-V
* BMI <17.5
* Patient attending an outpatient clinic at the Bohars Psychiatric Hospital in France
* Having signed the Informed Consent Form
* For minor patients, signing the form of informed consent of both parents

Exclusion Criteria:

* Associated eating disorder (bulimia, or the binge eating / purging form of anorexia nervosa),
* Psychiatric disorders (characterized depressed, anxiety disorder)
* Neurological Disorders
* Mental retardation
* Abuse or addiction to alcohol
* Abuse or dependence on psychoactive substances in the previous year.
* Patient with a protective justice measure

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Self-questionnaire assessing tolerance | Day 15
  Patients will have to respond to a self-administered questionnaire assessing tolerance
Self-questionnaire assessing acceptability | Day 15
  Patients will have to respond to a self-administered questionnaire assessing acceptability

SECONDARY OUTCOMES:
Feeling of presence | Day 15
  Patients will respond to a self-questionnaire of feeling of presence
Subjective experience by EDI-2 questionnaire | Day 15
  Pre- and post-test comparison of body dissatisfaction by EDI-2 questionnaire.
Subjective experience by BSQ questionnaire | Day 15
  Pre- and post-test comparison of body dissatisfaction by BSQ questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France